CLINICAL TRIAL: NCT01105195
Title: Efficacy of Surgical Preparations in Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: 3M (Industry)
Responsible Party: Michael Haak, MD, Northwestern University Feinberg School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00008875
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Infection
Keywords: DuraPrep; ChloraPrep; Lumbar Spine
MeSH Terms: conditions — Infections | interventions — DuraPrep

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DuraPrep (Active Comparator)
  Interventions: Other: DuraPrep
- ChloraPrep (Active Comparator)
  Interventions: Other: ChloraPrep

INTERVENTIONS:
Other: DuraPrep — DuraPrep is used for skin preparation prior to surgery.
  Arms: DuraPrep
Other: ChloraPrep — ChloraPrep is used for skin preparation prior to surgery.
  Arms: ChloraPrep

SUMMARY:
The purpose of this study is to 1) identify the common bacterial flora found on the skin overlying the lumbar spine, and 2) evaluate the efficacy of readily available skin-preparation solutions in the elimination of bacterial pathogens from the surgical site following skin preparation (DuraPrep versus ChloraPrep).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing lumbar spine surgery (discectomy, laminectomy, fusion, etc).

Exclusion Criteria:

* Open wound at the incision site,
* Abrasion in the vicinity of the incision site,
* An active infection at or near the surgical site, or
* An active infection elsewhere in the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Positive culture results | 7 days
  Our primary outcome measure is positive aerobic and/or anaerobic cultures reported at 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Background] Ostrander RV, Botte MJ, Brage ME. Efficacy of surgical preparation solutions in foot and ankle surgery. J Bone Joint Surg Am. 2005 May;87(5):980-5. doi: 10.2106/JBJS.D.01977. PMID 15866959
- See also: Information on ChloraPrep — http://www.chloraprep.com/
- See also: Information on DuraPrep — http://www.3m.com/product/information/DuraPrep-Surgical-Solution.html